CLINICAL TRIAL: NCT01241565
Title: A Prospective, Multi-Center Evaluation of the ENDO GIA™ Stapler With ENDO GIA™ Reload With Tri-Staple™ Technology in a Pulmonary Resection
Brief Title: ENDO GIA™ Stapler With ENDO GIA™ Reload With Tri-Staple™ Technology in a Pulmonary Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVEGTT0027
Record Dates: First submitted 2010-10-18; First posted 2010-11-16 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Lung Cancer
Keywords: lung cancer; lobectomy; wedge resection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ENDO GIA™ Stapler with TRI-STAPLE™ Technology (Experimental): Single arm study, all patients will receive the study device.
  Interventions: Device: ENDO GIA™ Stapler with TRI-STAPLE™ Technology

INTERVENTIONS:
Device: ENDO GIA™ Stapler with TRI-STAPLE™ Technology — All patients will have surgery with ENDO GIA™ Stapler with TRI-STAPLE™ Technology

SUMMARY:
The objectives of this clinical trial are to compare the incidence and duration of air leaks and the incidence of prolonged air leaks (defined as > 5 days by the Society for Thoracic Surgery) when using the ENDO GIA™ Stapler with ENDO GIA™ SULU with TRI-STAPLE™ Technology in a pulmonary resection via Video Assisted Thoracoscopic Surgery (VATS).

ELIGIBILITY:
Inclusion Criteria:

* The subject must be 18 years of age or older.
* The subject must be scheduled to undergo wedge resection or lobectomy via Video Assisted Thoracoscopic Surgery (VATS) for a lung nodule suspicious for or clinically proven to be primary lung cancer.
* The subject must be able to tolerate general anesthesia and have cardiopulmonary reserve to tolerate the procedure.
* The subject must be willing and able to comply with all study requirements and have understood and signed the informed consent.

Exclusion Criteria:

* The subject is pregnant or breastfeeding.
* The subject is scheduled to undergo sleeve lobectomy, segmentectomy, bi-lobectomy, pneumonectomy or Lung Volume Reduction Surgery (LVRS), or lung biopsy for suspected interstitial lung disease.
* A rib-spreading thoracotomy incision is scheduled to be performed, however the use of an access incision without rib-spreading for specimen removal or to facilitate hilar dissection is allowed. VATS procedures that are converted in the operating room to open procedures are not exclusionary.
* The subject has received pre-operative chemotherapy or radiation therapy for the lung cancer that will be resected.
* The subject is scheduled to receive intra-operative brachytherapy.
* The subject has other severe illnesses that would preclude surgery such as unstable angina or myocardial infarction within 3 months.
* Re-operative surgery is excluded if it is on the same side as the previous surgery.
* Investigator determines that participation in the study may jeopardize the safety or welfare of the subject.
* The subject is unable to comply with the follow-up visit schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert McKenna, MD, Principal Investigator — Cedar Sinai Medical Center
Locations (3):
- United States (3):
  - Cedar Sinai Medical Center, Los Angeles, California
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ENDO GIA™ Stapler With TRI-STAPLE™ Technology
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 128 subjects were screened for enrollment. 50 subjects were consented, enrolled and treated. There were 78 screen failures. 3 subjects were excluded from analysis, leaving 47 eligible subjects.
Arm/Group | ENDO GIA™ Stapler With TRI-STAPLE™ Technology
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (10.4)
Gender [Number; unit: participants]
  Female | 30
  Male | 17
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Prolonged Air Leaks
Description: Defined as > 5 days by the Society for Thoracic Surgery
Time Frame: Day 30
Measure: Number; unit: participants
Arm/Group | ENDO GIA™ Stapler With TRI-STAPLE™ Technology
Number analyzed (Participants) | 47
participants | 5
Statistical Analysis 1: Comparison: ENDO GIA™ Stapler With TRI-STAPLE™ Technology; Test type: Superiority or Other; Rate of incidence of PAL = 10.6, 95% CI 2-sided [3.9 to 21.3] — Incidence of Prolonged Air Leak (PAL) is estimated at between 5-10% in literature. PAL of 10%of evaluable cases was used to determine study success

2. Secondary Outcome: Incidence of Air Leaks
Description: As recorded on the air leak log.
Time Frame: Day 30
Measure: Number; unit: number of patients with air leaks
Arm/Group | ENDO GIA™ Stapler With TRI-STAPLE™ Technology
Number analyzed (Participants) | 47
number of patients with air leaks | 33

3. Secondary Outcome: Duration of Air Leak
Description: Measured in days. For patients discharged from the hospital with a Heimlich valve, the duration will be censored on the date of discharge.
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ENDO GIA™ Stapler With TRI-STAPLE™ Technology
Number analyzed (Participants) | 47
days | 3.52 (4.42)

4. Secondary Outcome: Length of Hospital Stay
Time Frame: Approximately Day 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ENDO GIA™ Stapler With TRI-STAPLE™ Technology
Number analyzed (Participants) | 47
days | 6.32 (5.59)

5. Secondary Outcome: Duration of Chest Tube Following Surgery
Description: Chest tube duration was calculated as removal date - placement date + 1
Time Frame: Approximately Day 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ENDO GIA™ Stapler With TRI-STAPLE™ Technology
Number analyzed (Participants) | 47
days | 5.02 (4.54)

6. Secondary Outcome: Incidence of Serosal Tearing
Time Frame: Day 30
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | ENDO GIA™ Stapler With TRI-STAPLE™ Technology
Number analyzed (Participants) | 47
participants | 2 [0.52 to 14.54]

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 30 days post surgery.
Arm/Group | ENDO GIA™ Stapler With TRI-STAPLE™ Technology
Serious Adverse Events (participants affected / at risk) | 10/47
Other Adverse Events (participants affected / at risk) | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENDO GIA™ Stapler With TRI-STAPLE™ Technology (N=47)
Atrial Fibrillation (Cardiac disorders) | 1 (1) — Atrial Fibrillation
Tachycardia (Cardiac disorders) | 1 (2) — Tachycardia
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1) — Mild Ischemic Colitis
Gastritis (Gastrointestinal disorders) | 1 (1) — Mild Gastritis
Pneumonia (Infections and infestations) | 1 (1) — Pneumonia
Tooth Abscess (Infections and infestations) | 1 (1) — Abscessed Tooth
Cerebrovascular Accident (Nervous system disorders) | 1 (1) — Stroke
Bronchopleural Fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Bronchopleural Fistula
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hemothorax
Hepatic Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hepatic Hydrothorax
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hypercapnia
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Aspiration Pneumonia
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Left Pneumothorax
Pulmonary Air Leakage (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Peristent Pulmonary Air Leak
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 2 (2) — Subcutaneous Emphysema
Hypotension (Vascular disorders) | 1 (1) — Hypotension
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENDO GIA™ Stapler With TRI-STAPLE™ Technology (N=47)
Cardiomegaly (Cardiac disorders) | 3 (3) — Cardiomegaly
Tachycardia (Cardiac disorders) | 3 (3) — Tachycardia
Urinary Tract Infection (Infections and infestations) | 3 (3) — Urinary Tract Infection
Incision Site Pain (Injury, poisoning and procedural complications) | 3 (3) — Incision Site Pain
Procedural Pain (Injury, poisoning and procedural complications) | 3 (4) — Procedural Pain
Neuralgia (Nervous system disorders) | 6 (6) — Neuralgia
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 28 (45) — Atelectasis
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) — Cough
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) — Dyspnea
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Hydropneumothorax
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Hypoxia
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 11 (14) — Lung Infiltration
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 11 (13) — Pleural Effusion
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 21 (23) — Pneumothorax
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 20 (21) — Subcutaneous Emphysema
Hypotension (Vascular disorders) | 3 (3) — Hypotension

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No